CLINICAL TRIAL: NCT06815666
Title: Prospective Study of Biomarkers Derived From Bronchoalveolar Lavage Fluid to Predict Outcomes in Soft-Tissue Sarcomas
Brief Title: BAL Fluid Biomarkers in Sarcoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-5871
Record Dates: First submitted 2025-01-26; First posted 2025-02-07 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Soft Tissue Sarcoma (STS); Bronchoalveolar Lavage (BAL); Bronchoalveolar Lavage Fluid
MeSH Terms: conditions — Sarcoma | interventions — Bronchoscopy; Metastasectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Routine Bronchoscopy & SOC Metastasectomy (Experimental): BALF and TA will be collected during routine bronchoscopy, and resected lung metastases and adjacent normal tissue will be collected during standard of care metastasectomy
  Interventions: Procedure: Bronchoscopy & Metastasectomy

INTERVENTIONS:
Procedure: Bronchoscopy & Metastasectomy — Routine bronchoscopy and standard of care metastasectomy

SUMMARY:
This is a single-centre, Phase II, prospective study designed to assess BALF and TA-derived biomarkers in relation to metastatic burden in STS patients. BALF and TA samples will be collected during routine bronchoscopy performed as part of standard care at Toronto General Hospital (TGH). Additionally, tissue samples of lung metastases and adjacent normal lung will be collected and used to correlate the identified biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Ability to understand and willingness to sign a written informed consent document
3. Diagnosed with soft tissue sarcoma
4. Undergoing resection of lung lesion as part of standard care

Exclusion Criteria:

1. History of another invasive malignancy, except for non-melanoma skin cancer or tumors curatively treated with no evidence of disease for ≥ 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2032-04-01 (Estimated); Study Completion 2032-04-01 (Estimated)

PRIMARY OUTCOMES:
Identification of NET-related inflammatory biomarkers using BALF and TA diagnostic tools | 2 years
  Bronchoalveolar lavage fluid (BALF) is a diagnostic tool used to sample cells and soluble substances from the lower respiratory tract. BALF allows for the examination of local immune responses and the identification of inflammatory markers. In the context of metastatic soft-tissue sarcoma, analyzing BALF can provide valuable insights into the presence and role of neutrophil extracellular traps (NETs) and other inflammatory factors within the lungs.
  On the other hand, tracheal aspirates (TA) can be more easily obtained from STS patients for biomarker identification.
Quantification of NET-related inflammatory biomarkers using BALF and TA diagnostic tool | 2 years
  Bronchoalveolar lavage fluid (BALF) is a diagnostic tool used to sample cells and soluble substances from the lower respiratory tract. BALF allows for the examination of local immune responses and the identification of inflammatory markers. In the context of metastatic soft-tissue sarcoma, analyzing BALF can provide valuable insights into the presence and role of neutrophil extracellular traps (NETs) and other inflammatory factors within the lungs.
  On the other hand, tracheal aspirates (TA) can be more easily obtained from STS patients for biomarker identification.
Correlation of NET-related inflammatory markers using BALF and TA diagnostic tool with the extent of metastatic dissemination | 2 years
  Bronchoalveolar lavage fluid (BALF) is a diagnostic tool used to sample cells and soluble substances from the lower respiratory tract. BALF allows for the examination of local immune responses and the identification of inflammatory markers. In the context of metastatic soft-tissue sarcoma, analyzing BALF can provide valuable insights into the presence and role of neutrophil extracellular traps (NETs) and other inflammatory factors within the lungs.
  On the other hand, tracheal aspirates (TA) can be more easily obtained from STS patients for biomarker identification.

SECONDARY OUTCOMES:
Analysis of NET-related inflammatory biomarkers using BALF and TA diagnostic tool | 2 years
  Comparative analysis of NET-related inflammatory biomarkers in BALF and tracheal aspirates. Collected specimens will undergo comprehensive multi-omic analysis, encompassing proteomic, transcriptomic, and DNA sequencing methodologies to characterize the molecular landscape of disease progression associated with NETs.
Correlation between NET-related inflammatory biomarkers using BALF and TA diagnostic tool | 2 years
  Correlation between the identified markers in BALF and tracheal aspirates with those found in resected pulmonary metastases and adjacent normal lung. The integration of these data will enable the identification of correlations between local and systemic disease features, uncovering potential biomarkers and pathways relevant to tumor progression and therapeutic targeting.
NET-related inflammatory biomarker differences for BALF and TA diagnostic tools | 2 years
  Assessment of any differences in NET-related inflammatory biomarker profiles between patients with different metastatic burdens. For BALF and TAs, the supernatant will be analyzed to identify inflammatory biomarkers and NET-associated proteins, while cellular components will be subjected to RNA sequencing for transcriptomic profiling and DNA sequencing to explore genetic and epigenetic modifications.

CONTACTS AND LOCATIONS:
Locations (1):
- Radiation Medicine Program, Princess Margaret Cancer Centre, University Health Network, Toronto, Ontario, Canada